CLINICAL TRIAL: NCT00246792
Title: Enhancing Self-Understanding and Social Integration of Middle School Students With Learning Disabilities
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); Integra LifeSciences Corporation (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14596
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2006-02-17 (Estimated); Status verified 2005-11

CONDITIONS: Learning Disability
Keywords: School-based intervention; Learning disabilities; ecological intervention
MeSH Terms: conditions — Learning Disabilities

INTERVENTIONS:
Behavioral: Group treatment

SUMMARY:
Research and intervention programs for students with learning disabilities (LD) typically address child and family characteristics without examining the school context and conditions that affect adjustment. Focusing on the student with LD can highlight the child and family's deficits. An ecological theoretical framework guides this research project, a collaboration of the University of Toronto, Faculty of Social Work and Ontario Institute for Studies in Education of the University of Toronto (OISE/UT), Integra and the Toronto Catholic District School Board. This framework is based on the assumption that people are very much part of and affected by social and environmental settings. Accordingly, it is important not to see the adjustment problems of children with LD as being caused only by their LD. Instead, their academic and social problems are seen as unfolding in larger circumstances that include other children, the classroom, the school, the family and the community. These many factors act together to influence the child with LD and must be taken into account along with individual characteristics of the child.

DETAILED DESCRIPTION:
Objectives

1. Deliver an ecologically informed school-based intervention that addresses individual, social and environmental factors, to improve the adjustment of students with LD
2. Examine the efficacy of the intervention
3. Contribute to knowledge of the factors that influence the adjustment of students with LD
4. Circulate this information to those who live and work with students with LD in order to offer understanding and direction for programs and interventions and to facilitate cross-sector collaboration

The research will utilize both quantitative and qualitative methodologies. 6 schools will be selected. 3 will receive the intervention in year 1 (2004-2005 school year), comprising 1) group treatment, 2) workshops, and 3) consultation. The other 3 schools will be controls in year 1 and receive the intervention in year 2 (2005-2006 school year).

Students in grades 6-8, identified as having LD will be offered the opportunity to participate in the project (with parental consent). This project comprises 3 components:

1. School-based group treatment for students in grades 6-8 with LD and psychosocial problems. Group treatment will focus on assisting participants to understand the impact of their LD as well as on development of self-advocacy skills.
2. Workshops on understanding LD for teachers, parents, and students without LD (grades 6-8).

ELIGIBILITY:
Inclusion Criteria:

* Grades 6-8 with identified LD
* Must demonstrate need for psychosocial intervention based on results on measures

Exclusion Criteria:

* Cannot meet criteria for conduct disorder on the Teacher Report Form

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2004-09; Study Completion 2006-12

PRIMARY OUTCOMES:
Child Behaviour Checklist (Achenbach, 2001)
Youth Report Form (Achenbach, 2001)
Teacher Report Form (Achenbach, 2001)

SECONDARY OUTCOMES:
Self-Perception Profile for Children (Harter, 1985)
The Children's Loneliness Questionnaire (Asher & Wheeler, 1985)
The Self Advocacy Interview for Students (Brunello-Prudencio, 2001)
Qualitative interviews with selected participants

CONTACTS AND LOCATIONS:
Overall Officials: Faye Mishna, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada